CLINICAL TRIAL: NCT07070375
Title: A Multicenter, Parallel-Group, Open-Label Study of Pharmacokinetics and Safety of HRS-8427 Injection in Chinese Subjects With Renal Impairment
Brief Title: Pharmacokinetics and Safety of HRS-8427 in Healthy Volunteers and in Patients With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8427-102
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gram-negative Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): Healthy volunteer with stable normal renal function
  Interventions: Drug: HRS-8427
- Cohort B (Experimental): Patient with stable mild renal impairment
  Interventions: Drug: HRS-8427
- Cohort C (Experimental): Patient with stable moderate renal impairment
  Interventions: Drug: HRS-8427
- Cohort D (Experimental): Patient with stable severe renal impairment
  Interventions: Drug: HRS-8427
- Cohort E (Experimental): Patient with end-stage renal failure.
  Interventions: Drug: HRS-8427

INTERVENTIONS:
Drug: HRS-8427 — HRS-8427

SUMMARY:
This study evaluated the pharmacokinetic profile, safety, and tolerability of HRS-8427 injection in subjects with mild, moderate, severe, or end-stage renal disease (ESRD) requiring dialysis, using subjects with normal renal function as controls, to inform clinical dosing in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 70 years old (including the boundary values);
2. The body weight of male subjects should be ≥ 50.0 kg, and that of female subjects should be ≥ 45.0 kg. The body mass index (BMI = body weight (kg) / height² (m²)) should be between 18.0 and 32.0 kg/m² (including the boundary values);
3. The estimated glomerular filtration rate (eGFR) (estimated by the MDRD formula) needs to meet the following criteria:

   For subjects with normal renal function: ≥ 90 mL/min and < 130 mL/min For subjects with mild renal insufficiency: 60 - 89 mL/min (including the boundary values) For subjects with moderate renal insufficiency: 30 - 59 mL/min (including the boundary values) For subjects with severe renal insufficiency: 15 - 29 mL/min (including the boundary values) For subjects with end-stage renal failure on maintenance dialysis: < 15 mL/min
4. The renal function status is stable. The interval between two detections during the screening period should be at least 72 hours (the result of the first detection can adopt the in-hospital or out-of-hospital detection result within 30 days before the second detection), and the absolute value of the fluctuation between the two detection results is less than 30%. Calculation formula: (the result of the second detection - the result of the first detection) / the result of the first detection;
5. Female subjects with fertility or male subjects whose partners are fertile females should have no plan for childbearing, donating sperm/eggs from the time of signing the informed consent form to 1 month after the last administration, and voluntarily take effective contraceptive measures (including partners) (non-drug contraception is required during the trial period).

Exclusion Criteria:

1. Subjects with a history of allergy to cephalosporins or penicillin, or those with specific allergic history (such as asthma, urticaria, eczema, etc.), or those with allergic constitution (such as being allergic to two or more drugs, foods and pollens);
2. Subjects who have undergone major surgeries within 3 months before screening, or those who have received surgeries that may significantly affect the in vivo process of the study drug or the evaluation of its safety, or those who plan to undergo surgeries during the trial period;
3. Subjects with a history of kidney transplantation or those who are expected to need kidney transplantation during the trial period;
4. Subjects who have been enrolled in any clinical trials as subjects within 3 months before screening;
5. Subjects with a positive result in any one of the tests for hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus (HIV) during the screening period;
6. From 48 hours before taking the study drug until the end of the study, subjects refuse to stop consuming any beverages or foods containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, grapefruit and beverages containing this ingredient, etc.);
7. Subjects who frequently drink alcohol within 6 months before screening (that is, female subjects who drink more than 14 standard units of alcohol per week, and male subjects who drink more than 21 standard units of alcohol per week (1 standard unit contains 14g of alcohol, such as 360 mL of beer or 45 mL of liquor with an alcohol content of 40% or 150 mL of wine)) or those who cannot refrain from drinking alcohol during the trial period;
8. Subjects with abnormal results of 12-lead electrocardiogram that are judged by the research doctor to be clinically significant or with a corrected QTcF ≥ 450 ms, etc.;
9. Subjects who cannot refrain from smoking during the trial period;
10. Subjects with a history of drug abuse/drug use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Cmax | 4 days
  observed maximum plasma concentration. Blood samples will be collected.
AUC0-t | 4 days
  area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected.
AUC0-∞ | 4 days
  area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected.
Tmax | 4 days
  observed time to reach Cmax. Blood samples will be collected.
Ae: amount excreted. Urine samples will be collected. | 4 days

SECONDARY OUTCOMES:
Incidence of treatment emergent AEs (TEAEs) | no more than 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided